CLINICAL TRIAL: NCT05229679
Title: Evaluation of Organized Human Papilloma Virus (HPV) Screening of 23-29-year-old Women
Brief Title: HPV-based Screening Among Women 23-29 Years of Age
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Joakim Dillner, Professor of Infectious Disease Epidemiology; Director of R&D, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-00053
Record Dates: First submitted 2021-11-30; First posted 2022-02-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Human Papilloma Virus; Cervical Intraepithelial Neoplasia; Cervical Cancer
Keywords: Organized screening; HPV vaccination; Human papilloma virus; Prevention
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV-based screening (Experimental): Women 23-29 invited to cervical screening will have their samples analyzed for HPV.
  Interventions: Diagnostic Test: HPV testing

INTERVENTIONS:
Diagnostic Test: HPV testing — All women age 23-29 resident in the pilot counties will be invited to HPV screening as of the study start date. The same invitation as currently used for women aged 30 and upwards will be used. This information clearly states that it is possible to opt out of the program and that data from the screening program will be collected to regional and national quality registers who will systematically evaluate the quality of the care. At the screening station, the samples are collected identically regardless of primary screening test used - there is no change in the procedures used neither for the woman or for the midwives taking the sample. HPV testing will be performed using the same purchased, CE-marked and accredited HPV screening platforms as currently used for women aged 30 and upwards. The cytology is according to the liquid-based cytology method.

SUMMARY:
The aim of the trial is to determine whether organized screening with primary HPV analysis provide higher cancer protection in the age group 23-29 years compared to primary cytology.

DETAILED DESCRIPTION:
The aim is to investigate whether primary HPV analysis in the organized cell sampling program for women in the age group 23-29 provides higher cancer protection compared to the current method where cell samples are primarily analyzed with cytology. In this study, all women in the age group 23-29 in the Stockholm and Skåne Region of Sweden will participate. Age is defined by year of birth. For 2020, women born 1991-1997 are included. Sampling and collection of samples is the same as for cytology.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 23-29 invited to screening.

Exclusion Criteria:

* Women who do not show up for screening or do not consent.

Ages: 23 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Individuals with a cervix and with a personal ID number indicating that they are a female, are eligible.
Enrollment: 180000 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2038-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of cervical cancer | Measured once during 1 year, year 1.
  Cervical cancer incidence in the intervention group compared to a historical control group.
Incidence of cervical cancer | Measured once during 1 year, year 2.
  Cervical cancer incidence in the intervention group compared to a historical control group.
Incidence of cervical cancer | Measured once during 1 year, year 3.
  Cervical cancer incidence in the intervention group compared to a historical control group.
Incidence of cervical cancer | Measured once during 1 year, year 4.
  Cervical cancer incidence in the intervention group compared to a historical control group.
Incidence of cervical cancer | Measured once during 1 year, year 5.
  Cervical cancer incidence in the intervention group compared to a historical control group.
Incidence of cervical cancer | Measured once during 1 year, year 6.
  Cervical cancer incidence in the intervention group compared to a historical control group.
Incidence of cervical cancer | Measured once during 1 year, year 7.
  Cervical cancer incidence in the intervention group compared to a historical control group.
Incidence of cervical cancer | Measured once during 1 year, year 8.
  Cervical cancer incidence in the intervention group compared to a historical control group.
Incidence of cervical cancer | Measured once during 1 year, year 9.
  Cervical cancer incidence in the intervention group compared to a historical control group.
Incidence of cervical cancer | Measured once during 1 year, year 10.
  Cervical cancer incidence in the intervention group compared to a historical control group.

SECONDARY OUTCOMES:
Cost-effectiveness of the new screening method | Measured once during 1 year, year 1.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.
Cost-effectiveness of the new screening method | Measured once during 1 year, year 2.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.
Cost-effectiveness of the new screening method | Measured once during 1 year, year 3.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.
Cost-effectiveness of the new screening method | Measured once during 1 year, year 4.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.
Cost-effectiveness of the new screening method | Measured once during 1 year, year 5.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.
Cost-effectiveness of the new screening method | Measured once during 1 year, year 6.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.
Cost-effectiveness of the new screening method | Measured once during 1 year, year 7.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.
Cost-effectiveness of the new screening method | Measured once during 1 year, year 8.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.
Cost-effectiveness of the new screening method | Measured once during 1 year, year 9.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.
Cost-effectiveness of the new screening method | Measured once during 1 year, year 10.
  Cost-effectiveness of HPV-based screening among women 23-29 as compared to cytology-based screening in the same age group. Cost data will be collected from the economy system used for the administration of the study, and compared to previous cost data.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Dillner, MD, PhD, Principal Investigator — Karolinska University Hospital/Karolinska Institutet
Locations (2):
- Sweden (2):
  - Region of Skåne, Lund, Skåne County
  - Region Stockholm, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
IPD has been discussed but a plan isn't finalized.